CLINICAL TRIAL: NCT03630081
Title: A Phase III, Randomized, Double-Blind, Multicenter, Comparative Study to Determine the Efficacy and Safety of Cefepime-Tazobactam vs. Meropenem Followed by Optional Oral Therapy in the Treatment of Complicated Urinary Tract Infection or Acute Pyelonephritis in Adults
Brief Title: Study of Cefepime-tazobactam (FEP-TAZ) in Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W-4282-301
Record Dates: First submitted 2018-07-23; First posted 2018-08-14 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: interventions — Meropenem; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WCK 4282 (FEP-TAZ) 4 g (Experimental): WCK 4282 (FEP-TAZ) Pharmaceutical dosage form: Intravenous infusion Dosage: 4 g (2 g FEP and 2 g TAZ) IV q8h, infused over 90 min
  Interventions: Drug: WCK 4282 (FEP-TAZ) 4 g; Drug: ciprofloxacin 500 mg Optional Oral Switch
- Meropenem (Active Comparator): Meropenem Pharmaceutical dosage form: Intravenous infusion Dosage: 1 g IV q8h, infused over 45 min
  Interventions: Drug: Meropenem; Drug: ciprofloxacin 500 mg Optional Oral Switch; Other: Infusion of normal saline

INTERVENTIONS:
Drug: WCK 4282 (FEP-TAZ) 4 g — WCK 4282 (FEP-TAZ) 4 g [2 g FEP and 2 g TAZ] IV q8h, infused over 90 min
  Arms: WCK 4282 (FEP-TAZ) 4 g
Drug: Meropenem — 1 g IV q8h, infused over 45 min
  Arms: Meropenem
Drug: ciprofloxacin 500 mg Optional Oral Switch — ciprofloxacin 500 mg PO q12h
Other: Infusion of normal saline — Infusion of normal saline over 45 min
  Arms: Meropenem

SUMMARY:
This is a Phase III, randomized, double-blind, multicenter, non-inferiority study to evaluate the efficacy, safety, and tolerability of FEP-TAZ vs. meropenem in the treatment of hospitalized adults with cUTI or AP.

DETAILED DESCRIPTION:
Approximately 1004 hospitalized adult subjects (≥18 years of age) diagnosed with cUTI or AP will be enrolled in the study. The diagnosis of cUTI or AP will be based on a combination of clinical symptoms and signs plus the presence of pyuria

Subjects will be randomized in a 1:1 ratio according to an Interactive Response Technology (IRT) electronic system to receive either FEP-TAZ 4 g (2 g cefepime + 2 g tazobactam) IV every eight hours (q8h) or meropenem 1 g IV q8h. FEP-TAZ will be administered as 2 consecutive infusions of 2 g (1 g cefepime + 1 g tazobactam)

ELIGIBILITY:
Inclusion Criteria:

Meet the following clinical criteria for either cUTI or AP:

A. cUTI:

1. Have at least TWO of the following new-onset or worsening symptoms or signs:

   Fever (oral, tympanic, or rectal temperature >38°C [>100.4°F]), which must be observed and documented by a health care provider Nausea or vomiting Dysuria, increased urinary frequency, or urinary urgency Lower abdominal, suprapubic, or pelvic pain
2. Have at least ONE complicating factor

B. AP, defined as acute flank pain (onset within 7 days prior to randomization) or costovertebral angle tenderness on physical examination, plus at least ONE of the following new-onset or worsening symptoms or signs:

3. Evidence of pyuria within 48 h prior to randomization,

Exclusion Criteria:

1. Known or suspected disease or condition that, in the opinion of the investigator, may confound the assessment of efficacy.
2. Receipt of potentially-effective systemic antibacterial therapy within 72 h prior to randomization
3. Rapidly progressive or terminal illness with a high risk of mortality due to any cause, including but not limited to acute hepatic failure, respiratory failure, or septic shock, such that the subject is unlikely to survive the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with overall success at Day 5 | Day 5
  Overall success is defined as complete resolution (or return to premorbid state) of the cUTI or AP symptoms that were present at screening, except flank pain (if present), which should show at least one grade improvement and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (reduced to <1000 colony forming units or CFU/mL)
Percentage of subjects with overall success at Test-of-Cure | Test Of Cure Visit (Day 17 ± 2 days)
  Overall success is defined as complete resolution1 (or return to premorbid state) of the cUTI or AP symptoms that were present at Screening and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (reduced to <1000 colony forming units or CFU/mL)
Percentage of subjects with Treatment-Emergent Adverse Events (TEAE) | Day 1 to the end of study Late Follow-Up visit (LFU) (26 ± 2 days)
  Collection of number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Manishkumar D Shah, PhD, Study Director — Wockhardt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isler B, Harris P, Stewart AG, Paterson DL. An update on cefepime and its future role in combination with novel beta-lactamase inhibitors for MDR Enterobacterales and Pseudomonas aeruginosa. J Antimicrob Chemother. 2021 Feb 11;76(3):550-560. doi: 10.1093/jac/dkaa511. PMID 33332545